CLINICAL TRIAL: NCT04686669
Title: A Phase 1, Randomised, Open-Label, Three-way, Three-period, Crossover Relative Bioavailability Study to Assess the Single-Dose Pharmacokinetics of FOR-6219 in Capsule and Tablet Formulations in Postmenopausal Women
Brief Title: A Relative Bioavailability Study of FOR-6219 in Capsule and Tablet Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forendo Pharma Ltd (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 40-533-002
Record Dates: First submitted 2020-12-11; First posted 2020-12-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Relative Bioavailability
Keywords: HSD17B1 inhibitor; Endometriosis; Food-effect; Bioavailability
MeSH Terms: conditions — Endometriosis | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Subjects receiving treatment sequence ABC (Experimental): Subjects will receive treatment sequence ABC on Days 1, 3 and 5 respectively; A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state, B= 3x50 milligrams FOR-6219 tablet given in fed state, C= 3x50 milligrams FOR-6219 tablet given in fasted state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation
- Subjects receiving treatment sequence BCA (Experimental): Subjects will receive treatment sequence BCA on Days 1, 3 and 5 respectively; B= 3x50 milligrams FOR-6219 tablet given in fed state, C= 3x50 milligrams FOR-6219 tablet given in fasted state, A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation
- Subjects receiving treatment sequence CAB (Experimental): Subjects will receive treatment sequence CAB on Days 1, 3 and 5 respectively; C= 3x50 milligrams FOR-6219 tablet given in fasted state, A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state, B= 3x50 milligrams FOR-6219 tablet given in fed state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation
- Subjects receiving treatment sequence ACB (Experimental): Subjects will receive treatment sequence ACB on Days 1, 3 and 5 respectively; A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state, C= 3x50 milligrams FOR-6219 tablet given in fasted state, B= 3x50 milligrams FOR-6219 tablet given in fed state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation
- Subjects receiving treatment sequence BAC (Experimental): Subjects will receive treatment sequence BAC on Days 1, 3 and 5 respectively; B= 3x50 milligrams FOR-6219 tablet given in fed state, A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state, C= 3x50 milligrams FOR-6219 tablet given in fasted state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation
- Subjects receiving treatment sequence CBA (Experimental): Subjects will receive treatment sequence CBA on Days 1, 3 and 5 respectively; C= 3x50 milligrams FOR-6219 tablet given in fasted state, B= 3x50 milligrams FOR-6219 tablet given in fed state, A= 3x50 milligrams FOR-6219 soft gelatine capsule given in fasted state.
  Interventions: Drug: FOR-6219 capsule formulation; Drug: FOR-6219 tablet formulation

INTERVENTIONS:
Drug: FOR-6219 capsule formulation — FOR-6219 capsule formulation will be available as a soft gelatine capsule with a single dose of 50 milligrams, administered orally.
Drug: FOR-6219 tablet formulation — FOR-6219 tablet formulation will be available as a tablet with a single dose of 50 milligrams, administered orally.

SUMMARY:
This is a phase 1, randomised, open-label, three-way, three-period, crossover relative bioavailability study to assess the single-dose pharmacokinetics of FOR-6219 in capsule and tablet formulations in postmenopausal women. The effect of high-fat food on the pharmacokinetics of the tablet formulation will also be evaluated. A total of twelve, post-menopausal women, will be randomised to receive a single oral dose of FOR-6219 in three treatment periods: capsule formulation (fasted); tablet formulation (fed); tablet formulation (fasted)

ELIGIBILITY:
Inclusion Criteria:

* Female participants between 45 and 65 years (inclusive) at screening
* Female participants must be either naturally (spontaneously) post-menopausal: Natural (spontaneous) postmenopause is defined as being amenorrheic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level >25.8 IU/L and 17β-oestradiol serum levels less than 183 pmol/L (or the local laboratory levels for post-menopause) OR Must have had a bilateral oophorectomy/bilateral salpingo-oophorectomy. Hysterectomised women can be included only if they have had bilateral oophorectomy.
* Participants not taking hormone replacement therapy (HRT).
* Has a body weight between 50kg and 100kg inclusive and a body mass index (BMI) between 18.5-30.0 kg/m^2 inclusive.
* Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation and urinalysis) that is reasonably likely to interfere with the participant's participation in or ability to complete the study as assessed by the investigator.
* Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any study-related procedures.
* Ability to swallow three capsules and tablets at a time or (consecutively) one capsule at a time.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Post-menopausal women with less than 12 months amenorrhoea, or women with amenorrhoea due to other medical causes.
* Current or recurrent disease (e.g., cardiovascular, haematological, neurological, endocrine, immunological, renal, hepatic or gastrointestinal or other conditions) that could affect the action, absorption, or disposition of FOR-6219, or could affect clinical laboratory evaluations.
* Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, use of prohibited therapies during the study or make the participant unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study may influence the result of the study, or the participant's ability to participate in the study.
* The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise-related clinically significant cardiac events.
* Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes.
* Has vital signs consistently outside of the following normal range. Supine blood pressure (after at least 5 minutes of supine rest): Systolic blood pressure: 90 - 140 mmHg, Diastolic blood pressure: 40 - 90 mmHg.
* Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
* Evidence of pregnancy
* Any other abnormal findings on vital signs, ECG, physical examination or laboratory evaluation of blood and urine samples that the Investigator judges as likely to interfere with the study or pose an additional risk in participating.
* Positive test results for alcohol or drugs of abuse.
* History or clinical evidence of substance and/or alcohol abuse within the two years before screening.
* Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within three months prior to the planned first day of dosing.
* Has used any medication that is either an inhibitor or inducer of CYP3A4 within 28 days or 10 half-lives (whichever is longer) prior to the planned first day of dosing. Additionally, participants must not have consumed other substances known to be potent inhibitors or inducers of cytochrome P450 (CYP P450s) in the two weeks before the planned first study drug administration.
* Has used any other prescription or over-the-counter medication (including herbal or homeopathic preparations; excluding vitamin/mineral supplements and occasional paracetamol) within 14 days or 10 half-lives (whichever is longer) prior to the planned first day of dosing that the Investigator judges is likely to interfere with the study or pose an additional risk in participating.
* Consumption of herbal remedies or dietary supplements containing St. John's Wort in the 3 weeks before the planned Day 1 of the dosing period.
* Has received an investigational product or been treated with an investigational device within 90 days prior to first drug administration and will not start any other investigational product or device study within 90 days after last study drug administration.
* Known or suspected intolerance or hypersensitivity to the investigational product, any closely related compound, or any of the stated ingredients.
* History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
* Has donated or lost 400 mL blood or more within the last 16 weeks preceding the first day of dosing.
* Has a mental incapacity or language barriers precluding adequate understanding, cooperation, and compliance with the study requirements.
* An inability to follow a standardised diet and meal schedule or inability to fast, as required during the study.
* Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomisation, participation, or enrolment in this study. Participants who initially failed due to temporary non-medically significant issues are eligible for rescreening once the cause has resolved.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Naturally (spontaneously) post-menopausal women or women with bilateral oophorectomy/bilateral salpingo-oophorectomy
Enrollment: 12 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Ratio of Peak Plasma Concentration (Cmax) after single dose of FOR-6219 tablet (fasted) over soft gelatine capsule (fasted) for FOR-6219. | Up to 48 hours postdose
Ratio of Area under the plasma concentration versus time curve (AUC) after single dose of FOR-6219 tablet (fasted) over soft gelatine capsule (fasted) for FOR-6219. | Up to 48 hours postdose
Ratio of Peak Plasma Concentration (Cmax) after single dose of FOR-6219 tablet (fed) over tablet (fasted) for FOR-6219. | Up to 48 hours postdose
Ratio of Area under the plasma concentration versus time curve (AUC) after single dose of FOR-6219 tablet (fed) over tablet (fasted) for FOR-6219. | Up to 48 hours postdose

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Time to peak plasma concentration (Tmax) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Terminal half-life (t½) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Area under the plasma concentration versus time curve (AUC) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Apparent total plasma clearance (CL/f) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Apparent volume of distribution during terminal phase (Vz/f) | Blood sampling up to the end of each treatment period: Up to 48 hours after the FOR-6219 dose in Period 1 and Period 2 and up to 96 hours after the FOR-6219 dose in Period 3
Incidence of Treatment Emergent Adverse Events (TEAE) | Adverse Events will be monitored from screening to 96 hours after the last FOR-6219 dose
Proportion of participants with morphological or rhythm abnormalities on Electrocardiograms (ECGs) | From Day -1 until 96 hours after the last FOR-6219 dose
  12-lead ECGs will be used to measure ECG
Proportion of participants with clinically significant changes in Electrocardiogram (ECG) PR time interval | From Day -1 until 96 hours after the last FOR-6219 dose
  12-lead ECGs will be used to measure ECG
Proportion of participants with clinically significant changes in Electrocardiogram (ECG) QRS time interval | From Day -1 until 96 hours after the last FOR-6219 dose
  12-lead ECGs will be used to measure ECG
Proportion of participants with clinically significant changes in Electrocardiogram (ECG) QT time interval | From Day -1 until 96 hours after the last FOR-6219 dose
  12-lead ECGs will be used to measure ECG
Proportion of participants with clinically significant changes in Electrocardiogram (ECG) QTc interval | From Day -1 until 96 hours after the last FOR-6219 dose
  12-lead ECGs will be used to measure ECG
Proportion of participants with clinically significant changes in laboratory safety tests | From Day -1 until 96 hours after the last FOR-6219 dose
  Laboratory safety tests include haematology, chemistry, coagulation and urinalysis
Proportion of participants with clinically significant changes in systolic blood pressure | From Day -1 until 96 hours after the last FOR-6219 dose
  Blood pressure will be measured using automated monitors in supine position after 5 minute rest.
Proportion of participants with clinically significant changes in diastolic blood pressure | From Day -1 until 96 hours after the last FOR-6219 dose
  Blood pressure will be measured using automated monitors in supine position after 5 minute rest.
Proportion of participants with clinically significant changes in pulse rate | From Day -1 until 96 hours after the last FOR-6219 dose
  Pulse rate will be measured using automated monitors in supine position after 5 minute rest.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, M.D., Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd., London, United Kingdom